CLINICAL TRIAL: NCT04190862
Title: An Open-Label, Single-Center, Investigator Initiated Phase 1B Trial of E-CEL UVEC as an Adjunct Cell Therapy for Treatment of Anal Fistulas
Brief Title: E-CEL UVEC as an Adjunct Cell Therapy for Treatment of Anal Fistulas
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Angiocrine Bioscience (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 19-04020122
Record Dates: First submitted 2019-12-05; First posted 2019-12-09 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Anal Fistula
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cell Therapy Treatment (Experimental): Patients who present with simple anal fistula and elect to undergo fistulotomy for treatment will be eligible to have E-CEL UVEC injected into the fistula at the time of fistulotomy to aid in healing.
  Interventions: Drug: E-CEL UVEC
- Cell Therapy Treatment Part BS1 (Experimental): Adult subjects with simple perianal fistula who meet all eligibility criteria to participate in Part B of the study will be treated in the outpatient setting with curettage and E-CEL UVEC cells without fistulotomy. E-CEL UVEC cells will be injected along the two sides (180 degrees apart from each other) of the whole length of the curetted anal fistula tract.
  Interventions: Drug: E-CEL UVEC
- Cell Therapy Treatment Part BS2 (Experimental): Subjects in Part B2-S will have the same eligibility criteria and would undergo the same procedure as described in Part B1, except that B2-S subjects will also have suturing and injection of the internal opening.
  Interventions: Drug: E-CEL UVEC
- Cell Therapy Treatment Part BM1 (Experimental): Subjects in Part BM1 will have the same eligibility criteria and would undergo the same procedure as described in Part B1, except that B2-M subjects in this cohort are eligible for up to 4 treatments (versus 1 in Part BS2).
  Interventions: Drug: E-CEL UVEC
- Cell Therapy Treatment Part BM2 (Experimental): This cohort comprises of multiple (M) treatments with E-CEL UVEC injections. The difference between Part BM1 and Part BM2, is that the subjects in the latter cohort receive double the dose of E-CEL UVEC cells per treatment. Subjects in Part BM2 will have the same eligibility criteria as Part BS1, BS2 and BM1 cohorts and would undergo the same treatment procedure as described in Parts BS1, BS2 and BM1.
  Every treatment consists of the percutaneous injection along both sides of the fistula tract plus injection of the internal opening via direct anoscopic visualization (described in the next paragraph). Dosing is 30 x 106 viable E-CEL UVEC cells into the area of the internal opening and minimum 30 x 106 viable E-CEL UVEC cells per centimeter along the fistula tract (15x106 viable E-CEL UVEC cells, each side per centimeter of the tract).
  All subjects in this cohort receive up to 6 treatments over 6 months. The six treatments are administered on visits WK 0, 3. 6, 9, 12 and 24.
  Interventions: Drug: E-CEL UVEC

INTERVENTIONS:
Drug: E-CEL UVEC — Injection of E-CEL UVEC

SUMMARY:
The purpose of this study is to determine if endothelial cells derived from human umbilical vein are safe for use in conjunction with fistulotomy for the treatment of simple anal fistulas. Endothelial cells are a special kind of cell in the body that line the inside surface of blood vessels. The goal of the study is to evaluate the preliminary safety of human umbilical vein cells in anal fistula healing.

DETAILED DESCRIPTION:
The purpose of this study is to test the safety of E-CEL UVEC® cells and see what effects (good and bad) it has on your anal fistula. It is hoped, that the E-CEL UVEC® cells may help to improve healing of your fistula after surgery.

E-CEL UVEC® cells are genetically engineered human endothelial cells that are taken from the umbilical cords of newborn babies. The endothelial cells are cells that line the inside of blood vessels including the umbilical cord. Human umbilical endothelial cells are collected from the umbilical cord of a healthy newborn baby. The cells are obtained under strict United States (U.S.) Food and Drug Administration (FDA) regulations. The endothelial cells are engineered in the laboratory, meaning an extra gene is added. A gene is taken from a virus (just a single gene, not the entire virus) and inserted into the endothelial cells.This causes the endothelial cells to be more stable and improves their growth capabilities. In animal studies, the endothelial cells were cleared from the body within a month. No negative side effects related to the endothelial cells were seen in animal studies. A higher than normal healing response was seen in animal studies.

This research study is being done because, in animal studies, E-CEL UVEC® cells have been shown to speed up healing in various tissues and organs. This study will test if it is safe to use E-CEL UVEC® cells and if they help to improve healing of your fistula after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subject ages 18 or older
* Subject willing and able to provide informed consent
* Subject is medically eligible and have agreed to undergo a fistulotomy
* Subject with simple perianal fistula with 2 or fewer fistula tracts
* Maximum tract length of 3 inches
* Subject without history of Crohn's disease/ Ulcerative Colitis
* For female subjects of childbearing potential:
* A negative serum or urine pregnancy test at screening is required prior to enrollment
* Subject must be willing to use a highly effective method of contraception from the start of the screening period throughout the study period
* For males who can father a child and are having intercourse with females of childbearing potential who are not using adequate contraception:
* Subject must be willing to use a recommended method of contraception and refrain from sperm donation from the start of the conditioning therapy for at least 1 year after completion and discussion with a treating physician

Exclusion Criteria:

* Concomitant rectovaginal fistulas
* Subjects with an abscess
* Presence of active infections findings (e.g.; redness, swelling, tenderness or fever)
* Presence of rectal and/or anal stenosis
* The presence of setons unless removed prior to the treatment
* Subjects with ongoing steroid treatment or treated with steroids in the last 4 weeks
* Renal impairment defined by creatinine clearance below 90 mL/min calculated using Cockcroft-Gault formula or by serum creatinine ≥ 1.5 x upper limit of normality (ULN)
* Hepatic impairment defined by both of the following laboratory ranges:
* Total bilirubin ≥ 1.5 x ULN unless benign congenital hyperbilirubinemia
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≥ 2.5 x ULN
* Known history of abuse of alcohol or other addictive substances in the 6 months prior to enrollment
* Active malignant tumor within 5 years
* Current recent history of abnormal, severe, progressive, uncontrolled hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurological, psychiatric, or cerebral diseases
* Congenital or acquired immunodeficiencies including human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS)
* Major surgery or severe trauma within the previous 6 months
* Subjects who are candidates for solid organ transplantation or who may have a high likelihood of needing a solid organ transplant (ex. progressive heart failure)
* Females who are who are pregnant or breastfeeding or planning to become pregnant or breastfeed during treatment
* Subjects who have known hypersensitivity or documented allergy to DMSO
* Subjects who do not wish to or cannot comply with study procedures
* Subjects currently receiving, or having received any investigational drug within 3 months prior to E-CEL UVEC cell therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2020-01-22 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2032-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety of dose escalation, as measured by incidence rate of treatment emergent adverse events following the administration of E-CEL UVEC | 2 weeks
  The short term safety of escalating dose of E-CEL UVEC cells in subjects with anal fistulas will be assessed by monitoring and recording all adverse events for 2 weeks following the administration of E-CEL UVEC. (Applicable to all arms)

SECONDARY OUTCOMES:
Efficacy of E-CEL UVEC, as measured the rate of subjects presenting with relapse in treated fistula | 6, 24 weeks after surgery
  Efficacy of E-CEL UVEC, as measured the rate of subjects presenting with relapse in treated fistula at week 6 and 24
  (Applicable to all arms)
E-CEL UVEC Treatment Success, as measured by the combination of cessation and absence of fistula leakage | 24 weeks after surgery
  The success of E-CEL UVEC cells in subjects with anal fistulas will be assessed via digital pressure after completion of all treatments.
  (Applicable to all arms)
Efficacy of E-CEL UVEC, as measured by time to complete healing of each side | 24 weeks after surgery
  Efficacy of E-CEL UVEC, as measured by time to complete healing of each side of injection site (Applicable to all arms)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey W Milsom, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College - NewYork-Presbyterian Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No